CLINICAL TRIAL: NCT06942936
Title: An Open-label, Fixed-sequence and Two-part Study to Assess the Impact of Multiple Doses of Itraconazole on the Pharmacokinetics of AZD5004 in Healthy Participants and Multiple Doses of AZD5004 on the Pharmacokinetics of Combined Oral Ethinyl Oestradiol and Levonorgestrel in Healthy Female Participants
Brief Title: A Study to Investigate the Impact of Multiple Doses of Itraconazole on AZD5004 in Healthy Participants and Multiple Doses of AZD5004 on Combined Oral Ethinyl Oestradiol and Levonorgestrel in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7260C00007; 2024-518467-35-00 (Other: EUCT number)
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: Part A and Part B are 2 independent and non-sequential parts (arms) in this study. Part A will be performed in healthy male and female participants. Part B will be performed in healthy female participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: AZD5004 + Itraconazole (Experimental): Participants will receive oral dose of AZD5004 on Period 1, followed by Itraconazole capsule orally in Period 2, and then will receive oral dose of AZD5004 combination with Itraconazole capsule in Period 3.
  Interventions: Drug: AZD5004; Drug: Itraconazole
- Part B: Ethinyl Estradiol/ Levonorgestrel (EE/LNG) + AZD5004 (Experimental): Participants will receive one tablet of combined 0.03/0.15 mg EE/LNG and AZD5004 orally.
  Interventions: Drug: AZD5004; Drug: EE/LNG

INTERVENTIONS:
Drug: AZD5004 — AZD50004 is administered orally as a tablet.
Drug: Itraconazole — Itraconazole is administered orally as a capsule.
  Arms: Part A: AZD5004 + Itraconazole
Drug: EE/LNG — EE/LNG is administered orally in the form of tablet.
  Arms: Part B: Ethinyl Estradiol/ Levonorgestrel (EE/LNG) + AZD5004

SUMMARY:
The purpose of this study is to assess the impact of multiple doses of itraconazole on the pharmacokinetics (PK) of AZD5004 in healthy participants (Part A), and to assess the impact of multiple doses of AZD5004 on the PK of Combined Oral Contraceptives (COCs) in healthy female participants (Part B).

DETAILED DESCRIPTION:
This study will be an open-label, fixed-sequence, two-part study in healthy participants.

There are 2 parts in this study:

Part A: performed in healthy male and female participants. Part B: performed in healthy female participants.

Part A will consist of:

1. Screening period of 27 days
2. Period 1
3. Period 2
4. Period 3
5. Follow-up period of 17 to 24 days after the last AZD5004 dose

Part B will consist of:

1. Screening period of 27 days
2. Start of study period
3. Up-titration period
4. End of study period
5. Follow-up

ELIGIBILITY:
Main Inclusion Criteria:

Part A -

* Suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of childbearing potential must not be lactating, must agree to use approved method of contraceptive.
* Sexually active fertile male participants with female partners of childbearing potential must adhere to the approved contraception methods.
* Have a Body Mass Index (BMI) between ≥ 18.5 kg/m2 and ≤ 35 kg/m2 (at the time of screening) and weigh at least 50 kg.

Part B -

* Females of non-childbearing potential must be confirmed at the Screening Visit by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhoea for at least 12 months following cessation of all exogenous hormonal treatments and Follicle-stimulating hormone (FSH) levels (> 40 mIU/mL).
  2. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation or tubal occlusion.
* Have a BMI between ≥ 23 kg/m2 and ≤ 30 kg/m2 and weigh at least 55 kg.

Main Exclusion Criteria:

Part A and Part B-

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study.
* History of acute pancreatitis (unless due to previously resolved gallstone pancreatitis and post-cholecystectomy), chronic pancreatitis, gallstones, or elevation in serum lipase/pancreatic amylase at screening.
* History or presence of any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Abnormal laboratory values, hepatic disease, Human Immunodeficiency Virus (HIV) positive, abnormal vital signs, abnormalities in rhythm, uncontrolled thyroid disease.
* Known smoker, history of alcohol, drug abuse or caffeine intake.
* Use of prescribed or unsubscribed medication within 3 months prior to screening.
* History of psychosis, bipolar disorder, major depressive disorder.
* Vulnerable participants, e.g., kept in detention, protected adults under guardianship.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Part A: Area under concentration-time curve from time zero to infinity (AUCinf) of AZD5004 | Day 1 and Day 10
  To assess the effect of multiple doses of itraconazole on the AUCinf of a single dose of AZD5004 in healthy male and female participants.
Part A: Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) of AZD5004 | Day 1 and Day 10
  To assess the effect of multiple doses of itraconazole on the AUClast of a single dose of AZD5004 in healthy male and female participants
Part A: Maximum observed drug concentration (Cmax) of AZD5004 | Day 1 and Day 10
  To assess the effect of multiple doses of itraconazole on the Cmax of a single dose of AZD5004 in healthy male and female participants
Part A: Terminal elimination half-life (t1/2λz) of AZD5004 | Day 1 and Day 10
  To assess the effect of multiple doses of itraconazole on the t1/2λz of a single dose of AZD5004 in healthy male and female participants
Part A: Time to reach maximum observed concentration (tmax) of AZD5004 | Day 1 and Day 10
  To assess the effect of multiple doses of itraconazole on the tmax of a single dose of AZD5004 in healthy male and female participants
Part A: Apparent total body clearance (CL/F) of AZD5004 | Day 1 and Day 10
  To assess the effect of multiple doses of itraconazole on the CL/F of a single dose of AZD5004 in healthy male and female participants
Part A: Apparent volume of distribution based on the terminal phase (Vz) of AZD5004 | Day 1 and Day 10
  To assess the effect of multiple doses of itraconazole on the Vz of a single dose of AZD5004 in healthy male and female participants
Part B: Area under concentration-time curve from time zero to infinity (AUCinf) of EE/LNG | Day 1, Day 8, Day 50 and Day 78
  To assess the effect of single and multiple oral dosing of AZD5004, at different dose levels of AZD5004, on the AUCinf of single doses of combined oral EE/LNG in healthy female participants
Part B: Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) of EE/LNG | Day 1, Day 8, Day 50 and Day 78
  To assess the effect of single and multiple oral dosing of AZD5004, at different dose levels of AZD5004, on the AUClast of single doses of combined oral EE/LNG in healthy female participants
Part B: Maximum observed drug concentration (Cmax) of EE/LNG | Day 1, Day 8, Day 50 and Day 78
  To assess the effect of single and multiple oral dosing of AZD5004, at different dose levels of AZD5004, on the Cmax of single doses of combined oral EE/LNG in healthy female participants
Part B: Terminal elimination half-life (t1/2λz) of EE/LNG | Day 1, Day 8, Day 50 and Day 78
  To assess the effect of single and multiple oral dosing of AZD5004, at different dose levels of AZD5004, on the t1/2λz of single doses of combined oral EE/LNG in healthy female participants
Part B: Time to reach maximum observed concentration (tmax) of EE/LNG | Day 1, Day 8, Day 50 and Day 78
  To assess the effect of single and multiple oral dosing of AZD5004, at different dose levels of AZD5004, on the tmax of single doses of combined oral EE/LNG in healthy female participants
Part B: Apparent total body clearance (CL/F) of EE/LNG | Day 1, Day 8, Day 50 and Day 78
  To assess the effect of single and multiple oral dosing of AZD5004, at different dose levels of AZD5004, on the CL/F of single doses of combined oral EE/LNG in healthy female participants
Part B: Apparent volume of distribution based on the terminal phase (Vz) of EE/LNG | Day 1, Day 8, Day 50 and Day 78
  To assess the effect of single and multiple oral dosing of AZD5004, at different dose levels of AZD5004, on the Vz of single doses of combined oral EE/LNG in healthy female participants

SECONDARY OUTCOMES:
Part A: Number of patients with Adverse Events (AEs) | From Screening (Day -2 to Day -28) to Day 27
  To assess the safety and tolerability of AZD5004 alone and in combination with itraconazole in healthy male and female participants
Part B: Number of patients with AEs | From Screening (Day -2 to Day -28) to Day 96
  To assess the safety and tolerability of AZD5004 alone and in combination with combined oral EE/LNG in healthy female participants
Part B: AUCinf of AZD5004 | Days 8, Day 50 and Day 78
  To assess the effect of single and multiple oral doses of AZD5004, at different dose levels of AZD5004, on the AUCinf of single doses of combined oral EE/LNG in healthy female participants.
Part B: AUClast of AZD5004 | Days 8, Day 50 and Day 78
  To assess the effect of single and multiple oral doses of AZD5004, at different dose levels of AZD5004, on the AUClast of single doses of combined oral EE/LNG in healthy female participants
Part B: Cmax of AZD5004 | Day 8, Day 50 and Day 78
  To assess the effect of single and multiple oral doses of AZD5004, at different dose levels of AZD5004, on the Cmax of single doses of combined oral EE/LNG in healthy female participants

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Baltimore, Maryland, United States
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/